CLINICAL TRIAL: NCT05075863
Title: Efficacy of Letrozole Versus Clomiphene Citrate on Ovulation Induction in Patients With Polycystic Ovarian Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nishtar Medical University (Other)
Responsible Party: Principal Investigator, Rashida Parveen, Consultant Gynecologist, Nishtar Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NishtarMU1
Record Dates: First submitted 2021-09-28; First posted 2021-10-13 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Letrozole

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clomiphene Citrate (Experimental): A total of 39 women were given clomiphene citrate, 100mg from 3 to 7 days of menstrual cycle. All patients underwent transvaginal scan (TVS) so that efficacy could be evaluated (ovulation occurs on 14 day of menstrual cycle after a treatment of 5 days of both groups. Induction of ovulation was assessed by TVS. If follicle of >2cm is found on 12 days TVS and smaller/collapsed on 16 days TVS, ovulation induction was labeled.
  Interventions: Drug: Letrozole
- Letrozole (Experimental): A total of 39 women were given letrozole, 5mg from day 3 to 7 of menstrual cycle. All patients underwent transvaginal scan (TVS) so that efficacy could be evaluated (ovulation occurs on 14 day of menstrual cycle after a treatment of 5 days of both groups. Induction of ovulation was assessed by TVS. If follicle of >2cm is found on 12 days TVS and smaller/collapsed on 16 days TVS, ovulation induction was labeled.
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole — Letrozole as 5mg from day 3 to 7 of menstrual cycle
  Other Names: Femara

SUMMARY:
We aimed this study to determine and compare frequency of induction of ovulation in women with polycystic ovarian syndrome treated with Letrozole versus clomiphene citrate as published literature shows variations.

DETAILED DESCRIPTION:
Discrepancy between ovulation induction rate and pregnancy rate is related to anti-estrogenic effects on cervical mucus and endometrium and long acting gonadotrophins are more effective than clomiphene citrate. This study was aimed at comparing frequency of induction of ovulation in women with polycystic ovarian syndrome treated with Letrozole versus clomiphene citrate.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed cases of polycystic ovarian syndrome.

Exclusion Criteria:

* All women having endocrine disorders like thyroid disorders.
* Women having hyperprolactinemia.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 78 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Induction of ovulation was assessed by Transvaginal scan (TVS) | 12 to 16 days.
  Induction of ovulation was assessed by TVS. If follicle of >2cm is found on 12 days TVS and smaller/collapsed on 16 days TVS, ovulation induction was labeled

CONTACTS AND LOCATIONS:
Overall Officials: Rashida Parveen, FCPS, Principal Investigator — Nishtar Medical University
Locations (1):
- Nishtar Medical University Hospital, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No